CLINICAL TRIAL: NCT04054752
Title: A Phase 1/1b Study of Enhancement of Immune Reconstitution and Vaccine Responses With Administration of Recombinant Human IL-7-hyFc (NT-I7) in Older Subjects Following Chemotherapy
Brief Title: Vaccine Response With NT-I7
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No subjects enrolled.
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NeoImmuneTech (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190134; 19-C-0134
Record Dates: First submitted 2019-08-10; First posted 2019-08-13 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Breast Carcinoma; Colorectal Adenocarcinoma; Bladder Carcinoma
Keywords: Breast Cancer; Colorectal Cancer; Immune Insufficiency; Bladder Cancer; Immunocompromised Host
MeSH Terms: conditions — Breast Neoplasms; Urinary Bladder Neoplasms; Colorectal Neoplasms | interventions — efineptakin alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/ Arm 1 (Experimental): NT-I7 administered at 720 and 960g/kg to select the OBD of NT-I7
  Interventions: Biological: Recombinant human IL-7-hyFc (NT-I7)
- 2/ Arm 2a (Active Comparator): Administration of 4 vaccines according to Sequence 1 + NT-I7 administration at OBD to assess vaccine response
  Interventions: Biological: Vaccine sequence 1
- 3/ Arm 2b (Active Comparator): Administration of 4 vaccines according to Sequence 2 + NT-I7 administration at OBD to assess vaccine response
  Interventions: Biological: Vaccine sequence 2

INTERVENTIONS:
Biological: Recombinant human IL-7-hyFc (NT-I7) — NT-I7 administered at escalating doses of 720, and 960g/kg to determine OBD of NT-I7
  Arms: 1/ Arm 1
Biological: Vaccine sequence 1 — Day 1 Immunization Pre-NT-I7:Td and Polio Day 64, Immunization Post-NT-I7: Hep A#1, Hep B#1 Day 106: Hep B#2 (Optional) 6 Month Post NT-I7 Vaccines (Optional): Polio, Hep A#2, Hep #3, PPSV23#1
  Arms: 2/ Arm 2a
Biological: Vaccine sequence 2 — Day 1 Immunization Pre-NT-I7: Hep A#1, Hep B#1 Day 64, Immunization Post-NT-I7:Td and Polio Day 106: no Vaccine 6 Month Post NT-I7 Vaccines (Optional): Polio, Hep A#2, Hep #3, PPSV23#1
  Arms: 3/ Arm 2b

SUMMARY:
Background:

People with cancer, and especially older people, have a weakened immune system (the defense system of the body). This is often caused by the treatments for cancer. Older cancer survivors are therefore more prone to getting infections, some of which are preventable through vaccines. But because their immune systems are weakened, their response to vaccines is poor. Researchers want to see if a new drug, NT-I7, can help.

Objective:

To see if NT-I7 can boost the immune system.

Eligibility:

Adults 60 and older who have recently finished chemotherapy for breast, colorectal, or bladder cancer.

Design:

Participants will be screened with a physical exam, medical history, and blood and urine samples. Their heart s electrical activity will be checked. They will have an ultrasound of their spleen. They may give a tissue sample from a previous biopsy.

Participants in phase 1a of the study will get 1 dose of NT-I7. It will be given by injection with a needle into the muscle of the upper arm, thigh, or buttocks.

Participants in phase 1b will get 5 vaccines over a few months. They may get an optional booster and/or 6th vaccine. They will also get NT-I7.

Participants will repeat the screening tests during the study. They may get a peripheral intravenous catheter in a vein in their hand or arm for blood draws.

Participants may have apheresis. For this, blood is taken from an arm vein. The white blood cells are separated from the blood. The rest of the blood, minus the white blood cells, is returned into a vein in the other arm. A catheter may be used.

Participants will have follow-up visits for 1 year.

DETAILED DESCRIPTION:
Background:

Interleukin-7 is a homeostatic cytokine with a critical role in lymphoid homeostasis through which it exerts its immune-restorative effects, particularly re-expansion of the na(SqrRoot) ve and memory T-cell subsets.

The clinical implications of the kinetics, nature and extent of immune reconstitution defects following standard or ablative chemotherapy in older adults with cancer (in particular the lack of reconstitution of large pools of na(SqrRoot) ve T-cell with broad repertoire diversity and of memory T-cells) are not well characterized.

As chemotherapy often induces only temporary complete or partial disease responses but no cure, candidates for novel immunotherapy strategies may be significantly impeded in their responses to active immunotherapy attempts, the therapeutic potential of which is becoming increasingly utilized.

Recombinant human IL-7 (rhIL-7) may play a role in immune reconstitution and immune enhancement in various circumstances of immune insufficiency in older individuals following chemotherapy or in the context of enhancing cancer immunotherapy or during immune senescence.

Elderly cancer survivors are vulnerable to vaccine-preventable diseases and are known to have poor anti-vaccine-specific immune responses. Effective prevention of communicable diseases is important for cancer survivorship.

This study will use NT-I7, a long acting IL-7 cytokine, composed of human IL-7 and a hybrid Fc (hyFc) region to extend half-life.

Objectives:

Phase 1: Select optimal biological dose (OBD) of NT-I7 in older subjects with breast, bladder, prostate or a gastrointestinal cancer following chemotherapy.

Phase 1b: Evaluate and quantify the functional impact of NT-I7 therapy on specific immune responses to selected vaccines in older subjects following chemotherapy.

Eligibility:

Adults greater than or equal to 60 year of age.

Diagnosis of non-metastatic breast, bladder or a gastrointestinal cancer following adjuvant / neo-adjuvant chemotherapy; or metastatic breast, gastrointestinal or prostate cancer after chemotherapy.

Completed a treatment with chemotherapy a minimum of 4 weeks and no more than 12 months prior to entry with no evidence of disease.

Reasonable expectation that no cancer-specific therapy will be given in the subsequent 6 months.

Design:

Subjects will be enrolled into this single center Phase 1/1b study following the specific therapy for their respective diseases.

In Phase 1 part of the study, two dose levels, 720 micro g/kg and 960 micro g/kg, will be compared. Six subjects will be enrolled in each dose level, and a single dose of NT-I7 will be delivered intramuscularly. The purpose of this part of the study is to select the OBD.

OBD is defined as the dose that yields the greatest rise in peak absolute total T-cell counts (peak value at any timepoint during the first 28 days post NT-I7 administration) with corresponding rise in na(SqrRoot) ve subsets of CD4+ and CD8+ T cells without accompanying substantial toxicities. Absolute increase is a delta between the baseline counts and the peak counts within each subject.

Once OBD is determined, the Phase 1b portion of this study will begin. Subjects will undergo immunizations with various antigens, randomized to be administered either before or after a single dose of NT-I7 at OBD. This inter-subject randomization of the order in which the immunizations are administered (according to the Sequence 1 or to the Sequence 2 schedule) will allow all immunocompromised subjects entered on the Phase 1b portion of the study to receive NT-I7.

The vaccines, randomly assigned to be administered before NT-I7 therapy are administered six weeks before the administration of NT-I7 therapy.

The vaccines, randomly assigned to be administered after NT-I7 therapy are administered 3 weeks after NT-I7 injection.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 60 years
* Documentation of positive diagnosis based on pathology/histology report (no need for archival tissue or new biopsy) for any of the following:

  * Stage I-III breast carcinoma following neo-adjuvant/adjuvant chemotherapy and appropriate surgery and/or radiotherapy.
  * Stage II or III gastrointestinal cancer following appropriate surgery and adjuvant chemotherapy or following appropriate neoadjuvant chemoradiation/surgery and adjuvant chemotherapy.
  * Stage II or III bladder carcinoma following neo-adjuvant chemotherapy and appropriate surgery or following adjuvant chemotherapy.
  * Stage IV breast, gastrointestinal, or prostate cancer, following surgery and chemotherapy, or chemotherapy alone

NOTE: "Appropriate therapy" for each disease must be consistent with NCCN Clinical Practice Guidelines in Oncology available at the time of treatment in the opinion of the investigator (http://www.nccn.org/professionals/physician_gls/f_guidelines.asp)

* Completed cancer specific therapy (including surgery, radiotherapy and/or systemic therapy) at least 4 weeks and no more than 12 months prior to registration. (Subjects with hormone receptor positive breast carcinoma maintained on hormonal therapy following chemotherapy and radiation are eligible. Subjects with HER2 positive breast carcinoma maintained on anti-HER2 agents after definitive therapies are also eligible).
* Reasonable expectation that no cancer-specific therapy, with the exception noted in the previous criteria, will be given in the subsequent 6 months (PI's discretion).
* Adequate organ function, as follows:

  * AST/ALT: < 3 times upper limit of normal (ULN)
  * Bilirubin: < 1.5 times ULN
  * Absolute Neutrophil Count: > 1000/mm3
  * Platelet count: > 75,000/mm3
  * INR/PTT: <1.5 times ULN
  * Serum Creatinine: <1.5 times ULN
  * CPK: <2.5 times ULN
  * Serum albumin: greater than or equal to 3g/dL
  * Serum electrolytes: within normal limits
* Karnofsky performance status greater or equal to 70%
* Effects of NT-I7 on the developing human fetus are unknown. For these reasons the following measures apply:

  * Subjects enrolled on the study must not be planning to father children within the projected duration of the trial, starting with the pre-screening/screening visit through 120 days after the administration of NT-I7.
  * Men with partners of childbearing potential (defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal (i.e., amenorrheic for greater than or equal to 12 months without alternative medical cause) must use effective contraception prior to study entry, and for 120 days after the administration of NT-I7.
  * Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, the study participants' treating physician should be informed immediately.

EXCLUSION CRITERIA:

* Subjects who are receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Significant heart disease defined as:

  * Significant coronary arterial disease
  * Myocardial infarction in the last 6 months, angina in the previous 3 months
  * Troponin elevation above reference range set by each institution where the troponin measurement was performed.
  * Ischemic changes on ECG
  * Atrio-ventricular block greater than 1st degree, in absence of pacemaker
  * QTc (using Fridericia and Framingham correction formula) greater than 480ms (CTCAE 5.0 grade 1 abnormality is acceptable)
  * History of ventricular arrhythmia
  * Left Ventricular Ejection Fraction of less than 50% determined by echocardiography
* Positive serology for HTLV-I or HIV, or serology findings indicative of ongoing infection with hepatitis A, hepatitis B, or hepatitis C. Subjects with serology findings indicative of previous exposure to hepatitis A or B vaccination will not be excluded from Phase 1 part of the study but will be excluded from Phase 1b part of the study (see below for additional exclusion criteria for the Phase-1b part of the study only).
* History of autoimmune disease EXCEPT for the following: subjects with vitiligo or endocrine disease controlled by replacement therapy including diabetes, thyroid, and adrenal disease may be enrolled
* Subjects requiring chronic immunosuppressive therapy (including corticosteroids above physiologic replacement dosage) for any medical condition. We will permit 1) systemic corticosteroids at physiologic replacement dosage which are not to exceed 10 mg/day of prednisone or an equivalent, 2) intranasal or inhaled corticosteroids, 3) intraarticular injection of corticosteroids, 4) topical corticosteroids, 5) or a short-term use of systemic corticosteroids greater than 10 mg/day of prednisone or an equivalent for 10 days or less.
* Splenomegaly or history of proliferative hematologic disease
* Prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation
* History of medical or psychiatric disease, or cognitive impairment, which, in the view of the principal investigator would preclude safe treatment
* Serious bleeding diathesis based on clinical history of significant bleeding attributed to coagulation/bleeding disorders, documentation of abnormal coagulation factors/platelet function studies at the discretion of PI, or those who are on therapeutic anticoagulation
* Inability to give informed consent
* Subjects who have received immune checkpoint inhibitors in the previous 12 months, or subjects who have received immunomodulatory drugs in the previous 4 weeks for any medical indications. Subjects who have received intravesical BCG administration for non-muscle invasive bladder cancer will be included in this study (i.e., not one of exclusion criteria).
* Additional exclusion criteria for the Phase-1b part of the study only are as follows:

  * Known hypersensitivity to any of the following: diphtheria toxoid, neomycin, polymixin B, streptomycin, 2 phenoxyethanol, formaldehyde, aluminum hydroxide, yeast
  * Previous exposure to Hepatitis A or B vaccines or history of hepatitis A or B infection
  * Subjects who received a Td or Tdap immunization in the previous 5 years
  * History of anaphylaxis or serious allergic reactions to previous administration of any of the vaccines
  * Subjects who had received one or more doses of the PPSV23 vaccine in the previous 12 months
  * Latex allergy
  * A history of Guillain-Barre syndrome within six weeks of administration of previous tetanus toxoid containing vaccines.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Phase 1: Safety of NT-I7 in elderly patients after chemotherapy | 28 days after treatment
  List of adverse events and frequency
Phase 1b: Evaluate and quantify if NT-I7 at optimal biological dose (OBD) has impacts on specific immune responses to vaccines | day 42 and day 106
  vaccine titers

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa A Hyder, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGAP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0134.html